CLINICAL TRIAL: NCT05401188
Title: Randomized Clinical Trial to Test the Efficacy and Safety of Outpatient Clinical Management of Urgent Laparoscopic Appendectomy in Uncomplicated Acute Appendicitis
Brief Title: Clinical Trial for a Outpatient Clinical Management of Urgent Laparoscopic Appendectomy
Acronym: ASI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HJ23 (Industry)
Collaborators: Hospital Universitari Joan XXIII de Tarragona. (Other)
Responsible Party: Principal Investigator, Jordi Elvira Lopez, Principal Investigator, HJ23
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2022-02-15; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Appendicitis Acute; Appendicitis
Keywords: outpatient management; Laparoscopic appendicectomy
MeSH Terms: conditions — Appendicitis | interventions — Hospitalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hospitalization group (Active Comparator): Patients in the hospitalization group, once the surgical intervention was finished, were transferred to the postoperative recovery unit and later they were discharged to the usual hospital ward. Patients received adequate intravenous fluid resuscitation based on their individual hemodynamic parameter and fluid balance, and they received analgesia according to personal requirement. In the hospital ward, the usual patient management protocols were followed until a complete recovery and consequently discharged according to the usual criteria.
  Interventions: Other: hospitalization
- outpatient group (Experimental): Patients in the outpatient group , once operated, were transferred to the surgery unit without admission and were later discharged home if they met the ALDRETE criteria in less than 23 hours after the intervention (following the surgery criteria without admission stages). If the patient was operated during the night shift, following the advice of major outpatient surgery where overnight stays are allowed, the patient was admitted to the post-anesthetic recovery unit and discharged the next day, always in less than 23 hours. In case of being discharged after 23 hours or not meeting ALDRETE criteria, it was considered a failure of the outpatient treatment.
  Interventions: Other: Outpatient

INTERVENTIONS:
Other: Outpatient — Once the patient was operated and an uncomplicated appendicitis was confirmed, the patient was randomized to one of the two experimental branches: the hospitalization group (HG) or outpatient group (OG). Patients in the OG were referred to the day-surgery unit where they were discharged according to ALDRETE criteria.
  Arms: outpatient group
Other: hospitalization — Once the patient was operated and an uncomplicated appendicitis was confirmed, the patient was randomized to one of the two experimental branches: the hospitalization group (HG) or outpatient group (OG). In this group, were admitted in the hospitalization ward.
  Arms: hospitalization group

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of outpatient management of uncomplicated acute appendicitis. For this purpose, a randomized clinical trial was designed. Selected patients who have undergone surgery for acute appendicitis are randomized into two groups. One group with hospitalization and another group without admission.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy and safety of outpatient management of laparoscopic appendicectomy in uncomplicated acute appendicitis.

This was a single center randomized controlled clinical trial consisting in 2 treatment groups. Patients were recruited in University Hospital of Tarragona Joan XXIII of Spain.

All patients admitted in the emergency department at University Hospital of Tarragona Joan XXIII with acute appendicitis diagnosis were likely to enter in the study. All patients who accomplished at least 4 over 5 of the Saint-Antoine criteria were included. The 5 criteria were: Leukocytosis lower than 15.000; C-Reactive protein lower than 30mg; Body mass index lower than 30kg/m2; appendicular diameter lower than 10mm and no radiological sign of complication.

All patients who met the inclusion criteria and none of the exclusion criteria were admitted to the study for emergency surgery.

In order to avoid the biases a unique anesthetic and surgical protocol were established for both groups.

Once Laparoscopic appendicectomy was performed the patients were randomly assigned to the hospitalization group or outpatient group.

Patients in the hospitalization group were admitted in the hospitalization ward. Patients in the outpatient group were referred to the day-surgery unit where they were discharged according to ALDRETE criteria.

The primary endpoint was the length of hospital stay (LHS). The length of hospital stay was calculated from the day and hour of admission in the surgical area to the day and hour of discharge, based on the hours of hospital stay. Secondary endpoints included the failures of the outpatient management, readmissions and the hospitals cost.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* meet at least 4 over 5 Saint Antoine criteria
* ASA classification (American Society of Anesthesiologists) less than or equal to 3
* patients who live accompanied in a home at a maximum distance of 30 minutes from the hospital and an adequate cognitive capacity.

Exclusion Criteria:

* pregnancy or breastfeeding
* complicated Acute Appendicitis
* surgical management performed in more 90 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — patients over 18 years old
Enrollment: 120 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
length of hospital stay (LHS) | up to 5 days
  The length of hospital stay (LHS) was calculated from the date and time of urgent appendectomy surgery to the date and time of hospital discharge, based on the hours of hospital stay (assessed up to 5 days)

SECONDARY OUTCOMES:
failures of the outpatient management | assessed up to 30 days
  Once the patients were discharged home, they were evaluated for emergency room visit. From the date of hospital discharge to the day of emergency room visit. The presence of a emergency room visit is considered as a Failure of the outpatient management.
readmissions | assessed up to 30 days
  Once the patients were discharged home, they were evaluated for readmission to the hospital ward. From the date of hospital discharge to the day of readmission to the hospital ward. The re-admission to the hospitalization ward was considered a readmission.
hospitals cost | through study completion, an average of 1 year
  The economic costs of both clinical managements were evaluated until the end of the study, a mean of 1 year. For the study, the direct and indirect costs of laparoscopic surgery, consumable material, economic expenses in the hospital ward, and the cost of the price of the emergency room visit were evaluated. The hospital's economic department was contacted and they calculated the cost in euros per patient. Each group was evaluated separately and a comparison was made.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Elvira Lopez, MD, Principal Investigator — HJ23
Locations (1):
- Jordi Elvira Lopez, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lefrancois M, Lefevre JH, Chafai N, Pitel S, Kerger L, Agostini J, Canard G, Tiret E. Management of Acute Appendicitis in Ambulatory Surgery: Is It Possible? How to Select Patients? Ann Surg. 2015 Jun;261(6):1167-72. doi: 10.1097/SLA.0000000000000795. PMID 24950287
- [Result] Paudel GR, Agrawal CS, Regmi R, Agrawal S. Conservative treatment in acute appendicitis. JNMA J Nepal Med Assoc. 2010 Oct-Dec;50(180):295-9. PMID 22049894
- [Result] Alvarado A. A practical score for the early diagnosis of acute appendicitis. Ann Emerg Med. 1986 May;15(5):557-64. doi: 10.1016/s0196-0644(86)80993-3. PMID 3963537
- [Result] Frazee RC, Roberts JW, Symmonds RE, Snyder SK, Hendricks JC, Smith RW, Custer MD 3rd, Harrison JB. A prospective randomized trial comparing open versus laparoscopic appendectomy. Ann Surg. 1994 Jun;219(6):725-8; discussion 728-31. doi: 10.1097/00000658-199406000-00017. PMID 8203983
- [Result] Cash CL, Frazee RC, Smith RW, Davis ML, Hendricks JC, Childs EW, Abernathy SW. Outpatient laparoscopic appendectomy for acute appendicitis. Am Surg. 2012 Feb;78(2):213-5. PMID 22369831
- [Result] Aubry A, Saget A, Manceau G, Faron M, Wagner M, Tresallet C, Riou B, Lucidarme O, le Sache F, Karoui M. Outpatient Appendectomy in an Emergency Outpatient Surgery Unit 24 h a Day: An Intention-to-Treat Analysis of 194 Patients. World J Surg. 2017 Oct;41(10):2471-2479. doi: 10.1007/s00268-017-4034-3. PMID 28474273
- [Result] Cash CL, Frazee RC, Abernathy SW, Childs EW, Davis ML, Hendricks JC, Smith RW. A prospective treatment protocol for outpatient laparoscopic appendectomy for acute appendicitis. J Am Coll Surg. 2012 Jul;215(1):101-5; discussion 105-6. doi: 10.1016/j.jamcollsurg.2012.02.024. Epub 2012 May 19. PMID 22609030
- [Result] Di Saverio S, Podda M, De Simone B, Ceresoli M, Augustin G, Gori A, Boermeester M, Sartelli M, Coccolini F, Tarasconi A, De' Angelis N, Weber DG, Tolonen M, Birindelli A, Biffl W, Moore EE, Kelly M, Soreide K, Kashuk J, Ten Broek R, Gomes CA, Sugrue M, Davies RJ, Damaskos D, Leppaniemi A, Kirkpatrick A, Peitzman AB, Fraga GP, Maier RV, Coimbra R, Chiarugi M, Sganga G, Pisanu A, De' Angelis GL, Tan E, Van Goor H, Pata F, Di Carlo I, Chiara O, Litvin A, Campanile FC, Sakakushev B, Tomadze G, Demetrashvili Z, Latifi R, Abu-Zidan F, Romeo O, Segovia-Lohse H, Baiocchi G, Costa D, Rizoli S, Balogh ZJ, Bendinelli C, Scalea T, Ivatury R, Velmahos G, Andersson R, Kluger Y, Ansaloni L, Catena F. Diagnosis and treatment of acute appendicitis: 2020 update of the WSES Jerusalem guidelines. World J Emerg Surg. 2020 Apr 15;15(1):27. doi: 10.1186/s13017-020-00306-3. PMID 32295644
- [Derived] Elvira Lopez J, Sales Mallafre R, Padilla Zegarra E, Carrillo Luna L, Ferreres Serafini J, Tully R, Memba Ikuga R, Jorba Martin R. Outpatient management of acute uncomplicated appendicitis after laparoscopic appendectomy: a randomized controlled trial. World J Emerg Surg. 2022 Nov 23;17(1):59. doi: 10.1186/s13017-022-00465-5. PMID 36419071